CLINICAL TRIAL: NCT00487383
Title: Suppression and Facilitation of the Motor Cortex by Stimulation of the Cerebellum in Patients With Dystonia and Healthy Controls
Brief Title: Brain Changes in Blepharospasm
Status: Terminated | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070165; 07-N-0165
Record Dates: First submitted 2007-06-15; First posted 2007-06-18 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2012-06-29

CONDITIONS: Dystonia; Focal Dystonia; Cerebellar Disease
Keywords: Cerebellum; Transcranial Magnetic Stimulation (TMS); Blepharospasm; DYT-1 Generalized Dystonia; Focal Dystonia; Dystonia; Healthy Volunteer; HV
MeSH Terms: conditions — Dystonia; Dystonic Disorders; Cerebellar Diseases; Blepharospasm

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will examine the role of certain areas of the brain in blepharospasm, a type of dystonia (abnormality of movement and muscle tone) that causes unwanted or uncontrollable blinking or closing of the eyelids. The study will compare brain activity in healthy volunteers and in people with blepharospasm to find differences in the brain that may lead to better treatments for dystonia.

Healthy volunteers and people with blepharospasm who are 18 years of age and older may be eligible for this study. All candidates are screened with a medical history. People with blepharospasm also have a physical examination and blepharospasm rating.

Participants undergo transcranial magnetic stimulation (TMS) and electromyography (EMG) in two 4-hour sessions, separated by 1 to 7 days.

TMS

A wire coil is held on the subject s scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. The subject hears a click and may feel a pulling sensation on the skin under the coil. There may be a twitch in muscles of the face, arm or leg. During the stimulation, subjects may be asked to tense certain muscles slightly or perform other simple actions. Repetitive TMS involves repeated magnetic pulses delivered in short bursts of impulses. Subjects receive 60 pulses per minute over 15 minutes.

EMG

Surface EMG is done during TMS to measure the electrical activity of muscles. For this test, electrodes (small metal disks) are filled with a conductive gel and taped to the skin of the face.

DETAILED DESCRIPTION:
Objective

Besides alterations in the basal ganglia, substantial evidence identifies cerebellar dysfunction as a possible cause for dystonia. Pathophysiological findings suggest that the cerebellar influence on the primary motor cortex is modified in patients with different forms of dystonia. The objective of this study is to find out whether this cerebellar influence plays a role in dystonic disorders.

Study population

20 patients with blepharospasm, 20 patients with focal hand dystonia, 20 patients with DYT-1 Primary generalized dystonia and 60 healthy volunteers age and sex matched.

Design

Paired pulse transcranial magnetic stimulation (TMS) will be performed at rest and during tonic activation of the first dorsal interosseus muscle (FDI). The conditioning stimulus (CS) will be applied to the ipsilateral cerebellum using different intensities and will precede the test stimulus by intervals from 3 to 10 ms, respectively. The test stimulus (TS) will be applied over the motor hot spot of FDI in the primary motor cortex.

Outcome measures

The primary outcome measure will be the motor evoked potential (MEP) in FDI after a conditioning cerebellar stimulus in relation to the unconditioned MEP size. Each different patient group will be compared separately to the age- and sex-matched healthy controls and between each other. Secondary outcome parameters will be the influence of different interstimulus intervals and different stimulation intensities of the conditioning stimulus on the MEP.

ELIGIBILITY:
* INCLUSION CRITERIA:

PATIENTS:

* Age 18 years or older
* Normal findings in the medical history, physical and neurological examination, except for dystonia

HEALTHY CONTROLS:

* Age 18 years or older
* Absence of dystonia or other neurological disorder with any effect on the motor or sensory systems

EXCLUSION CRITERIA:

Any of the following will exclude patients and controls from the study:

* Secondary forms of dystonia, including tardive dyskinesia
* History of seizure disorder
* Symptoms of a clinically relevant illness in the 2 weeks before the first study day, including history of any other neurological disorders or conditions requiring the use of anti-depressants, neuroleptic medications, anti-seizure medications, anticholinergic drugs, and muscle relaxants
* Taking the following medications: antidepressants, anxiolytics, anticonvulsants, antipsychotics, antiparkinson, hypnotics, stimulants, and/or antihistamines
* History of neuroleptic medications
* Presence of pacemaker, implanted medical pump, metal plate or metal object in skull or eye
* Botulinum toxin injection within 3 months of starting the protocol
* Known hearing loss

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-06-12; Study Completion 2012-06-29

CONTACTS AND LOCATIONS:
Overall Officials: Mark Hallett, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Albanese A, Barnes MP, Bhatia KP, Fernandez-Alvarez E, Filippini G, Gasser T, Krauss JK, Newton A, Rektor I, Savoiardo M, Valls-Sole J. A systematic review on the diagnosis and treatment of primary (idiopathic) dystonia and dystonia plus syndromes: report of an EFNS/MDS-ES Task Force. Eur J Neurol. 2006 May;13(5):433-44. doi: 10.1111/j.1468-1331.2006.01537.x. PMID 16722965
- [Background] Aramideh M, Koelman JH, Speelman JD, Ongerboer de Visser B. Eyelid movement disorders and electromyography. Lancet. 2001 Mar 10;357(9258):805-6. doi: 10.1016/s0140-6736(05)71235-6. No abstract available. PMID 11254003
- [Background] Aramideh M, Ongerboer de Visser BW, Holstege G, Majoie CB, Speelman JD. Blepharospasm in association with a lower pontine lesion. Neurology. 1996 Feb;46(2):476-8. doi: 10.1212/wnl.46.2.476. PMID 8614517